CLINICAL TRIAL: NCT04565392
Title: Proof-of-concept Randomized Placebo-controlled Trial of Famotidine for Outpatients With COVID-19
Brief Title: Remotely-conducted Trial of Famotidine vs Placebo for Patients at Home With Coronavirus (COVID) of 2019 (COVID-19)
Acronym: Pepcid4COV19
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: drpykessupplements.com (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pykonsult 201
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Covid19
Keywords: famotidine; Internet trial
MeSH Terms: conditions — COVID-19 | interventions — Famotidine

STUDY DESIGN:
Intervention Model Description: Parallel double-blind placebo-controlled interventional trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: study medication is Pepcid AC or matching placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- famotidine (Experimental): A 20-milligram tablet of Pepcid in the morning and evening the first day, to be increased thereafter to one tablet every 8 hours if not improving
  Interventions: Drug: Famotidine 20 milligram tablet
- Placebo (Placebo Comparator): A placebo tablet to match a 20-milligram (mg) tablet of Pepcid in the morning and evening the first day, to be increased thereafter to one tablet every 8 hours if not improving
  Interventions: Drug: Famotidine 20 milligram tablet

INTERVENTIONS:
Drug: Famotidine 20 milligram tablet — 1 tablet every 12 hours and increase to 1 tablet every 8 hours if not improved by the second day of treatment
  Other Names: Pepcid

SUMMARY:
Kit for reading vital signs (thermometer, wrist blood pressure device, finger oximeter) and with study drug is overnighted to qualified subjects with early symptoms of COVID-19. Subjects take a 20-milligram (mg) tab of famotidine or matching placebo twice a day, increase to 1 tablet every 8 hours if not better the 2nd day, and continue same for 30 days. Vital signs, symptoms, compliance etc are rechecked daily for the 30 days and once again 60 days after starting study drug. Consent, baseline, and follow-up are handled via internet plus calls/texts/virtual visits from study nurse or doctor as needed for clarifications and compliance.

DETAILED DESCRIPTION:
If an Over-The-Counter (OTC) medication could prevent worsening and hospitalization for COVID-19, it could stop the devastation wrought by the pandemic, and do so at a low cost. One OTC medication has a pre-clinical and clinical rationale to help: famotidine. For this study, 150 subjects are randomly assigned 50:50 to blinded treatment with 1 (20-milligram) tablet famotidine or matching placebo twice a day and can increase to 1 tablet three times a day. This internet-driven study requires subjects to maintain contact with and follow advice of their local MD, so it does not increase their risks from the disease. Baseline eligibility checklist follows informed consent. Subjects must have at least 5 of the standard symptoms of COVID19, be willing to keep taking study medicine and reporting results daily for 30 days, must start within the first 6 days of symptoms, and must have a study partner to complete their follow-up in case they become unable. The rate of subjects worsening or getting hospitalized is the main outcome measure.

ELIGIBILITY:
Inclusion Criteria:

1. - Probable COVID-19 based on presence of at least 5 of the following symptoms of acute onset within the prior 4 days: fever, cough, sore throat, fatigue, episodic chest pain or shortness of breath with exercise, muscle or body aches, headache, loss of smell or taste, stuffy or runny nose, chills or shivering, feeling hot or feverish, nausea, diarrhea
2. - Subjects must signify that they have contacted a doctor about their current symptoms.
3. - Subject gives informed consent for study and is willing to take the treatments and complete the scheduled evaluations.
4. - Subject has acquired a study partner who has agreed to complete the follow-up forms for the subject if the subject unable or has been hospitalized.

Exclusion Criteria:

1. - Constant rather than episodic trouble breathing, Persistent pain or pressure in the chest, New confusion, Inability to wake or stay awake, Bluish lips or face, or any other severe symptom [symptoms CDC urges immediate medical care for].
2. - Known sensitivity or intolerance to famotidine or another acid-blocking drug.
3. - Lack of access to the internet at home.
4. - Using tizanidine (Zanaflex® , a muscle relaxant), dasatinib (Sprycel®, a drug for leukemia), cefditoren (Pivoxil®, an antibiotic), or fosamprenavir or delavirdine (drugs for HIV) [Drug exclusions are per US label for Pepcid].
5. - Significant heart or kidney disease in the last 3 months according to subject's primary doctor
6. - Pregnant women
7. - Taking any investigational medications to treat COVID-19, famotidine, anti-viral drugs or corticosteroids and not stopping them within 48 hours before starting study treatment.

NOTE: patients are allowed to take over-the-counter agents for temporary relief of symptoms such as antipyretics and analgesics (aspirin, ibuprofen etc), cough remedies, anti-diarrheals, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Course Binary Outcome | 30th (last) day of treatment, or if discontinues treatment early, last observation carried forward
  Proportion of patients who self-rate as 6 on Patients Global Impression or are hospitalized for COVID-19 or similar symptoms or seek medical help for worsening symptoms, or get short of breath and have oxygen saturation below 90%, or die of COVID-19
Serious Adverse Events | 30th (last) day of treatment, or if discontinues treatment early, last observation carried forward]
  Proportion of patients who report a serious adverse event, i.e., one that causes hospitalization or death

SECONDARY OUTCOMES:
Time to symptomatic recovery | There is no baseline rating. Outcome is rated on the 30th (last) day of treatment, or if discontinues treatment early, last observation carried forward
  Proportion who answer the daily Global Recovery Question affirmatively: "Have you returned to your usual health (before your COVID-19 illness)? yes/no" if verified on the same day's evaluation by at least one category of improvement in each of the symptoms endorsed at baseline on the SCL18 (see Outcome 4).
SCL18 (self-check list of 18 symptoms of COVID-19) | Change from baseline at 30th (last) day of treatment, or if discontinues treatment early, last observation carried forward
  a) mean change in total (18-item) score since baseline; b) proportion self-rating each item (symptom) at a lower or 0 intensity value than at baseline; c) subtotal on: Major Acute Physical Symptoms (SCL18 #2, Pains in heart or chest, #4 Nausea, vomiting or upset stomach, #6 Sore throat, #7 Cough, #9 Chills or shivering, #11 Diarrhea, or #13, Trouble getting your breath), d) physical symptoms (first 13 items of SCL18), f) cognitive symptoms (last 5 items of SCL18). Each item is rated as (0) not at all, (1) a little bit (2) moderately, (3) quite a bit, or (4) extremely
Patient's Global Impression of Change | There is no rating at baseline. Outcome is for the 30th (last) day of treatment, or if discontinues treatment early, last observation carried forward
  Proportions rating Patient's Global Impression of Change: as 1-4; as 1-3; as 1-2; as 6 (answer set: 1, very much improved, 2/much improved, 3/moderately improved, 4/minimally improved, 5/about the same, 6/worse)
Adverse Events | 30th (last) day of treatment, or if discontinues treatment early, last observation carried forward
  Proportions of patients reporting new or worsening symptoms: a) any adverse event; b) the expected adverse events for famotidine (headache, dizziness, constipation, diarrhea); c) other adverse events, grouped by type
Day-60 Follow-up | 60 days after the start of treatment
  Each of the same endpoints as above but evaluated 30 days after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Pyke, MD, PhD, Principal Investigator — Pykonsult LLC
Locations (1):
- Pykonsult headquarters, New Fairfield, Connecticut, United States